CLINICAL TRIAL: NCT00209755
Title: Diagnostic Value of Plasma Ribavirin Assay During the Combination Therapy " Pegylated Interferon + Ribavirin " in Chronic Hepatitis C.
Brief Title: Plasma Ribavirin Assay During Combination Therapy for Chronic Hepatitis C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital A Michallon (Other)
Collaborators: University Hospital, Grenoble (Other); Central Hospital, Nancy, France (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ribatop - afssaps #031161
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2004-09

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

INTERVENTIONS:
Procedure: therapeutic drug monitoring of ribavirin and dose adaptation

SUMMARY:
Investigation of the usefullness of therapeutical drug monitoring of ribavirin for dose adaptation during combination therapy of chronic hepatitis C patients.

The correlation between ribavirin plasma concentration levels at week 4 (steady state) and early virological response (HCV-RNA decay from baseline to week 12) is to be tested in 40 patients approximately.

DETAILED DESCRIPTION:
1. Background and rational The serum concentrationS of ribavirin commonly range from 1 to 5 in patients during the combination treatment " interferon+ribavirin " (Larrat et al. 2003). However, the bioavailibility of ribavirin is not considered in the current recommendation for this treatment.

   The aim of this study is to demonstrate that the adaptation " à la carte " of ribavirin posology according to its serum concentration could improve the efficacy and the tolerance of the hepatitis C combination therapy.
2. Study design This study is a prospective clinical pharmacology trial in patients on combination treatment for a chronic hepatitis C with genotype 1 or 4 virus.

   The evaluation will concern the serum ribavirin concentration during the first three months of treatment and its correlation with the evolution of hemoglobin (toxicity marker) or viral load (efficacy marker).

   After the 3 months of the study, a adaptation of posology based on serum ribavirin level will be offer to the patients for the rest of the treatment period. A control of the ribavirin level one month after the dose adaptation will be performed.
3. Study treatments This trial is not a treatment evaluation. All the patients will receive the same treatment with PegInterferon alfa-2a and ribavirin according to the registered recommendations for use.
4. Target population The study population will consist of patients with genotype 1 or 4 chronic hepatitis C and for which a combination therapy is indicated.
5. Main selection criteria Patients with chronic hepatitis C related to genotype 1 or 4 virus and for which a combination therapy is needed will be eligible. Patients with co-infection (either VHB or VIH) or with concomitant treatments expected to interact with the endpoints (hemoglobin, viral load, serum ribavirin) will be excluded.
6. Judgement endpoints

   There will be intermediate endpoints :
   * blood hemoglobin concentration whom reduction during the 4 first weeks of treatment is a marker of toxicicty of the drug (induction of an hemolytic anemiae)
   * viral load whom reduction of at least 2 log after 12 weeks of treatment is correlated with the sustained virologic response to treatment
   * serum level of ribavirin for which it is expected a correlation with the two previous biological markers

   The primary judgement endpoint will be the statistical correlation as following :
   * the serum concentration of ribavirine at the plateau of pharmacokinetics (J28(S4))
   * the change of the hemoglobin concentration from D0 to D28(S4)
   * the change of hemoglobin concentration between D0 and D84(S12)
7. Secondary endpoints The thresholds of efficacy and toxicity of ribavirin will be determined by comparison of responder/non responder patients (as predicted by viral load change) and patients with/without toxicity. A correlation between the evolution of these two markers will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C related to genotype 1 or 4 virus and for which a combination therapy is needed will be eligible.

Exclusion Criteria:

* Patients with co-infection (either VHB or VIH) or with concomitant treatments expected to interact with the endpoints (hemoglobin, viral load, serum ribavirin) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Study Completion 2004-07

PRIMARY OUTCOMES:
relationship between plasma ribavirin concentration and early virological response

SECONDARY OUTCOMES:
safety
relationship between plasma ribavirin concentration and hemoglobin drop
dose effect of ribavirin on ribavirin plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre ZARSKI, MD, Principal Investigator — university hospital of Grenoble (France)
Locations (1):
- university hospital ; HGE dpt, Grenoble, France